CLINICAL TRIAL: NCT01380912
Title: Can Injection of Methylprednisoloneacetate 80 mg, in the Cavity After Mastectomy for Primary Breast Cancer, at the Time of Removal of the Drain, Prevent Seroma Formation?
Brief Title: Can Methylprednisoloneacetate Prevent Seroma After Mastectomy for Primary Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Charlotte Lanng, MD, Department of Breast Surgery ,Herlev Hospital
Other Study IDs: H-4-2009-137
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; mastectomy; methylprednisoloneacetate; seroma; numbers of punctures
MeSH Terms: conditions — Breast Neoplasms; Seroma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — seroma will be analysed for concentration of cytokines, and eventual growth of bacteria
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- breast cancer: 1. Patients operated with mastectomy and axillary dissection, who are randomised to injection of methylprednisoloneacetate in the cavity
  2. Patients operated with mastectomy and axillary dissection, who are randomised to injection of saline solution in the cavity
  3. Patients operated with mastectomy and Sentinel Node Operation, who are randomised to injection of methylprednisoloneacetate in the cavity
  4. Patients operated with mastectomy and Sentinel Node Operation, who are randomised to injection of saline solution in the cavity
  Interventions: Drug: methylprednisoloneacetate

INTERVENTIONS:
Drug: methylprednisoloneacetate — Either methylprednisoloneacetate 80 mg or saline solution will be injected first day after operation, when the drain is removed.

SUMMARY:
A randomised double-blinded study, in which the patients either get methylprednisoloneacetate or saline solution in the mastectomy cavity to evaluate the efficacy of methylprednisoloneacetate in preventing seroma in patients operated for primary breast cancer.

DETAILED DESCRIPTION:
After mastectomy, up to 90 % of patients develops seroma in the cavity. The treatment is puncture, which is a small operation, but many patients have to come several times, and there is a risk of infection. In some cases further treatment can be postponed.

Preventing seroma to develop would be an improvement in the treatment of breast cancer patients operated with mastectomy.

An earlier study found that the seroma production was significant lower in the group who had Prednison injected directly into the cavity.

In this study the patient are divided into two groups: patients who have mastectomy and axillary dissection and patients who have mastectomy and Sentinel Node operation. Each group are examined separately.

Using Prednison in patients after operation could be a potential risk, but correct injection into the cavity will seldom give systemic side effects.

ELIGIBILITY:
Inclusion Criteria:

* women with primary breast cancer or Ductal carcinoma in situ, mastectomy plus either Sentinel Node or Axillary dissection, signed consent form

Exclusion Criteria:

* dissection of the axilla in les than 4 month, treatment with steroids, pregnancy, if the patient don't speak danish, allergy towards steroid, other medical conditions which the investigator find contradict participating

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for primary breast cancer with mastectomy and eihter axillary dissection or Sentinel Node operation
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
number of punctures | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gro M Qvamme, MD, Principal Investigator
Locations (2):
- Denmark (2):
  - Chemistry Laboratorium, Copenhagen University Hospital at Gentofte, Hellerup
  - Department of Breast Surgery, Copenhagen University Hospital at Herlev, Herlev